CLINICAL TRIAL: NCT00302328
Title: A Randomised Clinical Trial of Prognostic Factors and Surgical Methods for the Treatment of Idiopathic Macular Holes
Brief Title: Trial of Prognostic Factors and Surgical Methods for the Treatment of Idiopathic Macular Holes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Collaborators: Danish Eye Health Society (Other); The Danish Medical Research Council (Other)
Responsible Party: Principal Investigator, Ulrik Christensen, MD, Glostrup University Hospital, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COMAH
Record Dates: First submitted 2006-03-13; First posted 2006-03-14 (Estimated); Results first posted 2014-04-16 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-03

CONDITIONS: Idiopathic Macular Hole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- macular hole operation no peeling (No Intervention)
- Macular hole operation ICG peeling (Active Comparator)
  Interventions: Procedure: macular hole operation
- Macular hole operation TB peeling (Experimental)
  Interventions: Procedure: macular hole operation

INTERVENTIONS:
Procedure: macular hole operation — macular hole surgery with either no peeling, indocyanine green (ICG) assisted peeling or trypan blue (tb) peeling
  Arms: Macular hole operation ICG peeling; Macular hole operation TB peeling

SUMMARY:
The project is a randomized clinical trial with a follow up time of 12 months comparing the effects of surgical treatment of idiopathic macular holes. Patients are randomized to vitrectomy alone, vitrectomy plus indocyanine green (ICG) assisted inner limiting membrane ( ILM) peeling or vitrectomy plus trypan blue (tb) assisted ILM peeling. At baseline patients are characterized using early treatment diabetic retinopathy study (ETDRS) visual charts, tests of aniseikonia, optical coherence tomography 3 (OCT3), visual field and fundus photography. Per- and postoperative complications are registered.

Data analyses will help clarify the effect of ILM peeling on hole closure and visual acuity. Comparing results after ICG- and tb assisted ILM peeling will help clarify the topic of a toxic effect on retinal cells after staining and peeling of the ILM. Changes in intraretinal morphology before and after dye-assisted ILM peeling will be studied using OCT3 imaging and the patients' subjective opinion on the surgical results will be analyzed using quality of life questionnaires and metamorphopsia tests.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic macular hele stage 2 or 3.
* Duration of Symptoms ≤ 12 months.
* Visual acuity ≥ 34 ETDRS letters.
* Intraocular pressure ≤ 23 mmHg.
* Informed consent.

Exclusion Criteria:

* Previous macular hole in project eye
* Macular pucker worse than a cellophane macular reflex.
* Previous surgery or disease in the eye affecting retinal function.
* Systemic disease affection vision including diabetes mellitus with level of retinopathy ≥ 14a.
* Amblyopia i project eye.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2005-08; Primary Completion 2008-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Morten la Cour, MD,DMSc,EBOD, Study Director — Glostrup Hospital, Department of Ophthalmology; Michael Larsen, MD, DMSc, Study Director — Glostrup Hospital, Department of Ophthalmology
Locations (1):
- Department of Ophthalmology, Glostrup Hospital, Copenhagen, Denmark

REFERENCES:
- [Derived] Christensen UC. Value of internal limiting membrane peeling in surgery for idiopathic macular hole and the correlation between function and retinal morphology. Acta Ophthalmol. 2009 Dec;87 Thesis 2:1-23. doi: 10.1111/j.1755-3768.2009.01777.x. PMID 19912135
- [Derived] Christensen UC, Kroyer K, Sander B, Jorgensen TM, Larsen M, la Cour M. Macular morphology and visual acuity after macular hole surgery with or without internal limiting membrane peeling. Br J Ophthalmol. 2010 Jan;94(1):41-7. doi: 10.1136/bjo.2009.159582. Epub 2009 Aug 18. PMID 19692379
- [Derived] Kroyer K, Christensen U, la Cour M, Larsen M. Metamorphopsia assessment before and after vitrectomy for macular hole. Invest Ophthalmol Vis Sci. 2009 Dec;50(12):5511-5. doi: 10.1167/iovs.09-3530. Epub 2009 Jul 2. PMID 19578018
- [Derived] Christensen UC, Kroyer K, Sander B, Larsen M, Henning V, Villumsen J, la Cour M. Value of internal limiting membrane peeling in surgery for idiopathic macular hole stage 2 and 3: a randomised clinical trial. Br J Ophthalmol. 2009 Aug;93(8):1005-15. doi: 10.1136/bjo.2008.151266. Epub 2008 Nov 21. PMID 19028741
- [Derived] Kroyer K, Christensen U, Larsen M, la Cour M. Quantification of metamorphopsia in patients with macular hole. Invest Ophthalmol Vis Sci. 2008 Sep;49(9):3741-6. doi: 10.1167/iovs.07-1452. Epub 2008 Apr 30. PMID 18450594

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 3 years
Groups:
- no Peeling: no peeling used
- ICG Peeling: indocyanine (ICG) peeling
- tb Peeling: trypan blue (tb) peeling
Period: Overall Study
Arm/Group | no Peeling | ICG Peeling | tb Peeling
Started | 25 | 35 | 18
Completed | 25 | 34 (developed cancer during the study) | 18
Not Completed | 0 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- ICG Peeling: indocyanine green (ICG) peeling
- Total: Total of all reporting groups
Arm/Group | no Peeling | ICG Peeling | tb Peeling | Total
Number analyzed (Participants) | 25 | 35 | 18 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 25 | 10 | 50
  >=65 years | 10 | 10 | 8 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.6 (5) | 66.9 (5) | 66.6 (5) | 66.6 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 27 | 9 | 56
  Male | 5 | 8 | 9 | 22
Region of Enrollment [Number; unit: participants]
  Denmark | 25 | 35 | 18 | 78

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity (ETDRS Letters)
Description: Visual acuity measured as the number of ETDRS letters at last follow-up
Time Frame: Visual acuity at 12 months
Population: Decided from initial power calculation
Measure: Mean (Standard Error); unit: Visual acuity in letters
Groups:
- no Peeling: Vitrectomy without peeling
- ICG Peeling: vitrectomy with icg-assisted ilm peeling
- tb Peeling: vitrectomy with trypan blue assisted ilm peeling
Arm/Group | no Peeling | ICG Peeling | tb Peeling
Number analyzed (Participants) | 25 | 34 | 18
Visual acuity in letters | 74.9 (8.2) | 72.4 (6.5) | 72.2 (9.1)

2. Secondary Outcome: Anatomic Success
Description: closure of the macular hole evaluated on optical coherence tomography 3 (OCT3)
Time Frame: macular hole closure at 12 months
Population: from initial power calculation of primary end point
Measure: Number; unit: participants
Groups:
- no Peeling: vitrectomy without ilm peeling
- ICG Peeling: vitrectomy with icg assited ilm peeling
- tb Peeling: vitrectomy with trypan blue assited ilm peeling
Arm/Group | no Peeling | ICG Peeling | tb Peeling
Number analyzed (Participants) | 25 | 34 | 18
participants | 11 (31) | 32 | 16

3. Secondary Outcome: Visual Field Defects
Description: visual field defects measured on humphrey perimetry
Time Frame: 6 months
Population: from predetermined power analysis
Measure: Number; unit: participants
Arm/Group | no Peeling | ICG Peeling | tb Peeling
Number analyzed (Participants) | 25 | 34 | 18
participants | 0 [0 to .1] | 1 | 1

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | no Peeling | ICG Peeling | tb Peeling
Serious Adverse Events (participants affected / at risk) | 14/25 | 3/35 | 2/18
Other Adverse Events (participants affected / at risk) | 0/25 | 0/35 | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | no Peeling (N=25) | ICG Peeling (N=35) | tb Peeling (N=18)
cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
macular hole did not close (Eye disorders) | 14 | 2 | 2

LIMITATIONS AND CAVEATS:
non-closure of macular hole after surgical procedure in 18 patients led to re-operation. Data included in main published papers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No